CLINICAL TRIAL: NCT01257958
Title: Vitamin D Pilot Study in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: HSC #97-676-311
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Vitamin D, 19 nor Vitamin D, Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 19 nor vitamin d (Experimental)
  Interventions: Drug: 19 nor vitamin d

INTERVENTIONS:
Drug: 19 nor vitamin d

SUMMARY:
Phase 1 study of 19-nor Vitamin D in relapsing-remitting MS. Primary measure is MRI.

ELIGIBILITY:
Inclusion Criteria:

* relapsing remitting MS

Exclusion Criteria:

* MRI contraindicated

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-02; Primary Completion 2000-02 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
MRI Measure of new active lesions, observation vs. treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UW-Madison, Madison, Wisconsin, United States